CLINICAL TRIAL: NCT07098611
Title: A New Tool for Extubation Readiness in Mechanically Ventilated Patients: Readiness for EXtubation Score (REXs STUDY)
Brief Title: A New Tool for Extubation Readiness in Mechanically Ventilated Patients: Readiness for EXtubation Score
Acronym: REXs
Status: Recruiting | Type: Observational
Sponsor: Medipol University (Other)
Collaborators: International Association of Non Invasive Ventilation (Unknown); International Academy of Non Invasive Ventilation (Unknown); International College of Experts of Non Invasive Ventilation (Unknown)
Responsible Party: Principal Investigator, Berkan Basançelebi, Lecturer, Medipol University
Other Study IDs: IRB00010984
Record Dates: First submitted 2025-07-19; First posted 2025-08-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ventilator Weaning; Respiration, Artificial; Respiratory Failure; Extubation Readiness; Extubation Failure; Extubation Succeeded; Intensive Care Patients Invasively Ventilated; Weaning Invasive Mechanical Ventilation
Keywords: mechanical ventilation; extubation; weaning; readiness; prediction; score
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing weaning from invasive mechanical ventilation: In patients who are prepared for extubation, predictive readiness will be assessed with REXs.

SUMMARY:
Liberation from mechanical ventilation involves three steps: weaning, readiness assessment, and extubation. Readiness is determined using clinical criteria such as improvement of the underlying condition, hemodynamic stability, and adequate respiratory effort. Successful extubation is defined as not requiring invasive support within 48 hours. Due to the complexity of ICU patients, various clinical parameters and multi-component scores have been developed to predict extubation success. This study aims to develop and evaluate a multi-component score, the Readiness for EXtubation score (REXs), to predict extubation readiness in ICU patients under invasive mechanical ventilation.

DETAILED DESCRIPTION:
Background: Liberation from mechanical ventilation (MV) involves a three-step process; weaning, readiness testing, and extubation. Readiness testing uses objective clinical criteria to determine whether a patient is ready to begin weaning from MV. These criteria include improvement of the underlying indication for MV, hemodynamic stability, and the ability to initiate and sustain both adequate inspiration and expiration. Successfully extubation from invasive MV is a critical milestone in the recovery from severe respiratory failure and and is a clinical challenge for clinicians.

Spontaneous breathing trials (SBT) are conducted to evaluate a patient's readiness for ventilator liberation in the intensive care unit (ICU). Extubation is considered successful if invasive mechanical support is not required within 48 hours after the removal of the endotracheal tube. As the final step of the weaning process, the decision to extubate is typically guided by objective criteria demonstrating the patient's ability to sustain respiratory function without mechanical assistance. Considering the complex pathologies of intensive care patients, besides SBT many clinical parameters have been used as predictors of weaning and extubation. For this reason, different multi-component scales and scores have been developed.

The study protocol is designed and will be reported in accordance with the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement.

The aim of this study is to develop a multi-component Readiness for EXtubation score (REXs) that can predict extubation readiness and to analyze this score that can be applied to patients under invasive MV in the ICU.

Sample Size: The sample size was calculated as 427 using the Area Under ROC Curve in the ExPreS study. The total targeted sample size was accepted 470 patients with estimating that there would be a 10% dropout.

Screening and Admission: The daily screen will be performed between 8:00 and 10:00 a.m. by the clinician assigned to the unit each morning that the patient was on invasive mechanical ventilation. Patients meeting the criteria will be included in the study.

Data Collection and Anonymization: The data collected are part of routine clinical care, and the data will be anonymized. Clinicians will add anonymously the data they obtain to a created electronic case report form (e-CRF). Clinicians will be allowed to assign numbers to patients so that they can be distinguished by the clinicians who add them.

The dataset that constitute the e-CRF for each patient are; demographics (country, age, sex, BMI), ICU type, cause of ICU admission, number of comorbidities, weaning/extubation type, SBT duration, arterial blood gases (ABG: pH, PaCO2, PaO2), ventilation parameters (brand/model, FiO2, PEEP, ventilation index, RSBI, MVspont/MVtotal, PCF, P0.1, vital capacity, NIF, Cdyn), secretion type, agitation and sedation score (RASS), heart rate, hemoglobin, nutrition target percentage, ventilatory support after extubation, extubation failure (24,48 and 72 hrs), duration of invasive MV, ICU and hospital length of stay and mortality.

pH: It measures the acidity or alkalinity of blood and is crucial for assessing acid-base balance. Normal arterial pH is 7.35-7.45. A pH lower than 7.35 indicates acidosis, while a pH higher than 7.45 indicates alkalosis. Abnormal pH can indicate metabolic or respiratory disorders. The pH of the blood is crucial when assessing the success of weaning. The pH outside the normal range can indicate an imbalance in acid-base homeostasis, which may suggest inadequate respiratory function or metabolic disturbances that would make weaning unsafe. Maintaining a normal pH ensures that the patient's respiratory and metabolic systems can function without requiring excessive ventilatory support.

PaCO2: PaCO2 is a direct measure of ventilation. During weaning, a PaCO2 level within normal limits is needed for extubation success. Persistent hypercapnia during weaning suggests that the patient may be unable to sustain adequate ventilation on their own, leading to potential failure.

PaO2/FiO2: This ratio is a measure of the severity of hypoxemia. During weaning, a higher PaO2/FiO2 ratio suggests that the lungs are functioning well enough to support breathing without mechanical assistance. A low ratio suggests the need for continued mechanical ventilation.

PEEP: PEEP is used to prevent alveolar collapse and improve oxygenation. When weaning, reducing PEEP gradually helps assess whether the patient can maintain oxygenation without it. High levels of PEEP might be detrimental when reducing ventilatory support, as it can affect weaning success.

Ventilation Index (VI): The ventilation index (VI) combines respiratory rate and tidal volume, giving an overall assessment of ventilation efficiency. A low VI is favorable during weaning because it indicates that the patient is able to achieve adequate ventilation with minimal support. VI is calculated as VI="(PIP* PaCO2*RR)/1000".

Rapid Shallow Breathing Index (RSBI): The rapid shallow breathing index (RSBI), also known as the ratio of respiratory rate to tidal volume (RR/VT), is the most commonly used predictor of weaning success due to its simplicity and ease of interpretation. The clinical utility of the RSBI is emphasized in the 2007 international consensus guidelines for weaning from mechanical ventilation, the 2007 Brazilian consensus guidelines, and the 2013 Brazilian guidelines for mechanical ventilation, all of which recommend its use.

MVspont/MVtotal: This ratio reflects the proportion of ventilation that is spontaneous versus mechanical in one minute. A higher spontaneous ventilation (MVspont) relative to total ventilation (MVtotal) indicates that the patient is relying less on mechanical support, which may be reflect favorable for weaning.

Peak Cough Flow (PCF): PCF is an indicator of a patient's ability to clear secretions. Secretion retention is a key factor in weaning failure, as it increases respiratory load and is often linked to an ineffective cough. Evaluating cough strength in ICU patients can help predict weaning outcomes, as insufficient cough strength appears to be associated with higher in-hospital mortality. Consequently, assessing cough strength in intubated patients is increasingly being integrated into ICU extubation protocols. The subject is instructed to take a deep breath and cough as forcefully as possible. The clinician then freezes the ventilator screen and measures the maximal expiratory flow (L/min) from the flow curve. Clinicians can use the mechanical ventilator's algorithm if available. The average of three successful measurements will be taken.

P0.1: In a study on healthy subjects, Whitelaw et al. conducted random, brief end-expiratory occlusions using a specialized circuit during both resting and CO2 rebreathing. They observed that the decrease in airway pressure (Paw) within the first 100 milliseconds (0.1 s) of an occluded breath remained relatively constant, was consistent for each subject under different conditions, and correlated more strongly with end-tidal CO2 than with minute ventilation. They introduced this parameter as airway occlusion pressure Pocc, or P0.1. P0.1 reflects the inspiratory effort of the patient. It is used to assess the respiratory drive. Normal P0.1 suggests that the patient has adequate respiratory drive to maintain spontaneous breathing. Clinicians can use the mechanical ventilator's algorithm if available. The average of three successful measurements will be taken.

Vital Capacity (VC): Vital capacity (VC) reflects the total volume of air a person can exhale after a maximal inhalation. During weaning, a VC of at least 10-15 mL/kg is generally considered adequate for successful extubation. Vital capacity is measured by instructing patients to inhale deeply to their maximum capacity, followed by a forceful exhalation. The clinician then freezes the ventilator screen and measures maximal volume (mL) from the volume curve. Clinicians can use the mechanical ventilator's algorithm if available. The maximum of three successful measurements will be taken.

Negative Inspiratory Force (NIF): Negative inspiratory force (NIF), also referred to as maximum inspiratory pressure, reflects the maximal effort of the inspiratory muscles during inhalation against an obstructed airway. This index is used to evaluate respiratory muscle strength, with a value greater than - 30 cm H2O serving as a criterion for initiating the mechanical ventilator weaning process. After exhaling, the patient is given the command to take a deep breath. The clinician freezes the screen when the patient perform the fastest inhalation during expiratory hold maneuver. The clinician measures the minimum pressure from the pressure curve. Clinicians can use the mechanical ventilator's algorithm if available. The minimum of three successful measurements will be taken.

Cdyn: Dynamic compliance is a measure of lung and chest wall compliance during mechanical ventilation. High compliance typically indicates less stiff lungs, which is favorable during weaning. It is obtained by dividing the VT by the difference between PIP and PEEP.

Secretion: In mechanically ventilated patients, the primary mechanisms of secretion clearance-mucociliary transport and cough-are impaired. Major contributing factors to pulmonary secretion retention include the presence of an artificial airway, insufficient humidification of inspired gases, and limited mobility. Ineffective secretion clearance increases the risk of ventilator dependency and reintubation due to airway obstruction, aspiration, or infection.

Agitation/Sedation: Effective management of agitation and sedation is essential for successful weaning in mechanically ventilated patients, as both excessive sedation and agitation can impede the process. Over-sedation reduces respiratory drive, weakens respiratory muscles, prolongs ventilation, and increases the risk of ventilator-associated pneumonia. In contrast, agitation can heighten the work of breathing, increase the risk of self-extubation, and cause cardiovascular strain. The Richmond Agitation-Sedation Scale (RASS) is a 10-point tool that categorizes patient states, ranging from severe agitation (+4, combative) to deep sedation and unresponsiveness (-5), with 0 indicating a calm and alert state.

Heart rate: Heart rate is an important indicator of cardiovascular stability during weaning. A significant increase in heart rate during mechanical ventilation or SBTs can signal distress, leading to the suspension of the weaning attempt.

Hemoglobin: The impact of hemoglobin levels on weaning outcomes in mechanically ventilated patients remains controversial, with limited data, particularly for those experiencing difficult weaning. Patients with weaning difficulties may benefit more from higher hemoglobin levels than those in the early stages of respiratory failure, as sufficient hemoglobin is essential for adequate oxygen delivery during the weaning process. Lower hemoglobin levels reduce arterial oxygen content, impair oxygen delivery, and increase respiratory muscle workload, potentially hindering successful weaning.

%Nutrition Target: Adequate nutrition is essential for survival and reducing hospital stay in critically ill patients, as it supports muscle strength, including respiratory muscles, which is crucial for successful weaning from mechanical ventilation. Malnutrition can impair weaning by weakening respiratory function. To guide evidence-based nutritional therapy, several global guidelines have been published. The American Society for Parenteral and Enteral Nutrition (ASPEN) and the Society of Critical Care Medicine (SCCM) recommend energy intake of 25-30 kcal/kg/day and protein intake of 1.2-2.0 g/kg/day, while the European Society for Parenteral and Enteral Nutrition (ESPEN) suggests 20-25 kcal/kg/day with 1.3 g/kg of protein equivalents per day.

Statistical Analysis: Statistical analysis will be performed using IBM SPSS Statistics 26 (IBM Corp., Armonk, NY, USA). Categorical variables will be summarized as numbers (n) and frequencies (%). The Fisher's exact test will be applied for 2×2 contingency tables, and the Chi-square test will be used for all other contingencies to evaluate associations between clinical/demographic characteristics and extubation success or failure. For continuous variables, the Shapiro-Wilk test will be used to assess normality of distribution. Normally distributed variables will be summarized as means (± standard deviation), while non-normally distributed variables will be expressed as medians (with interquartile range). The independent samples Student's t-test will be employed to compare groups for normally distributed variables, and the Mann-Whitney U test will be used for non-normally distributed variables. All parameters with a p-value < 0.4 in group comparisons (extubation success vs. failure) will be further investigated using univariable logistic regression analysis to assess their association with extubation outcome; odds ratios (OR) and 95% confidence intervals (CI) will be calculated. Receiver operating characteristic (ROC) analysis will be performed to evaluate the predictive value of each parameter. The cutoff values optimizing sensitivity and specificity will be determined using the Youden Index. The REXs cutoffs used in comparisons will be established based on the Youden Index. Finally, REXs cutoff values indicating low, moderate, and high probability of extubation risk will be determined.

ELIGIBILITY:
Inclusion Criteria:

- Patients who are in the weaning process from mechanical ventilation after being connected to invasive mechanical ventilation in the intensive care unit.

Exclusion Criteria:

* Patients without legal guardian consent.
* Tracheostomized patients.
* Patients enrolled in other studies.
* Individuals with diaphragmatic pacers.
* Pregnant patients.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on mechanical ventilation admitted to the Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Extubation failure in 48 hours | From the beginning of the extubation process until 48 hours after extubation
  Extubation failure within 48 hours is defined as the need for reintubation or resumption of mechanical ventilation within two days after planned extubation, indicating the patient could not sustain spontaneous breathing independently.

SECONDARY OUTCOMES:
Extubation failure in 72 hours | From the beginning of the extubation process until 72 hours after extubation
  Extubation failure within 72 hours is defined as the need for reintubation or resumption of mechanical ventilation within three days after planned extubation, indicating the patient could not sustain spontaneous breathing independently.
Extubation failure in 24 hours | From the time of extubation until 24 hours post-extubation.
  Patients included who present failure in extubation from mechanical ventilation in the first 24 hours post extubation and require orotracheal intubation
Length of intensive care stay | From admission to intensive care to discharge
  Length of intensive care stay refers to the total number of days a patient spends in the intensive care unit (ICU) from admission to discharge, reflecting the severity of illness and recovery progress.
Length of hospital stay | From admission to hospital to discharge
  Length of hospital stay (LOS) refers to the total number of days a patient remains admitted in the hospital from initial admission until final discharge, serving as an important indicator of treatment efficiency and healthcare resource utilization.
Intensive care mortality | From admission to intensive care to discharge
  Intensive care mortality refers to the proportion of patients who die during their stay in the intensive care unit (ICU), serving as a critical indicator of ICU performance and patient outcomes.
Hospital mortality | From admission to hospital to discharge
  Hospital mortality refers to the proportion of patients who die during their hospitalization, from admission to discharge, serving as a key indicator of healthcare quality and patient outcomes.

CONTACTS AND LOCATIONS:
Locations (7):
- University of Magallanes, Punta Arenas, Chile
- Cairo University, Cairo, Egypt
- Shahid Beheshti University of Medical Sciences, Tehran, Iran
- Italy (2):
  - A.O.R.N. "Dei Colli" Monaldi Hospital, Napoli
  - Monaldi-Cotugno Hospital, Napoli
- Hospital General Universitario Morales Meseguer, Murcia, Spain
- İstanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
During the publication phase of the study, all data will be anonymized and made available as supplementary material accompanying the published article.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Result] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Result] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Result] Lai YC, Ruan SY, Huang CT, Kuo PH, Yu CJ. Hemoglobin levels and weaning outcome of mechanical ventilation in difficult-to-wean patients: a retrospective cohort study. PLoS One. 2013 Aug 28;8(8):e73743. doi: 10.1371/journal.pone.0073743. eCollection 2013. PMID 24015310
- [Result] da Silva RB, Neves VR, Montarroyos UR, Silveira MS, Sobral Filho DC. Heart rate variability as a predictor of mechanical ventilation weaning outcomes. Heart Lung. 2023 May-Jun;59:33-36. doi: 10.1016/j.hrtlng.2023.01.007. Epub 2023 Jan 26. PMID 36706686
- [Result] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Result] Volpe MS, Guimaraes FS, Morais CC. Airway Clearance Techniques for Mechanically Ventilated Patients: Insights for Optimization. Respir Care. 2020 Aug;65(8):1174-1188. doi: 10.4187/respcare.07904. PMID 32712584
- [Result] Ghiani A, Walcher S, Lutfi A, Gernhold L, Feige SF, Neurohr C. Mechanical power density, spontaneous breathing indexes, and weaning readiness following prolonged mechanical ventilation. Respir Med. 2025 Feb;237:107943. doi: 10.1016/j.rmed.2025.107943. Epub 2025 Jan 7. PMID 39788438
- [Result] Vu PH, Tran VD, Duong MC, Cong QT, Nguyen T. Predictive value of the negative inspiratory force index as a predictor of weaning success: a crosssectional study. Acute Crit Care. 2020 Nov;35(4):279-285. doi: 10.4266/acc.2020.00598. Epub 2020 Nov 30. PMID 33423439
- [Result] Korupolu R, Uhlig-Reche H, Achilike EC, Reeh C, Pedroza C, Stampas A. Factors Associated With Ventilator Weaning Success and Failure in People With Spinal Cord Injury in an Acute Inpatient Rehabilitation Setting: A Retrospective Study. Top Spinal Cord Inj Rehabil. 2022 Spring;28(2):129-138. doi: 10.46292/sci21-00062. Epub 2022 Apr 12. PMID 35521063
- [Result] Macnaughton PD. Assessment of lung function in the ventilated patient. Intensive Care Med. 1997 Aug;23(8):810-8. doi: 10.1007/s001340050417. No abstract available. PMID 9310798
- [Result] Whitelaw WA, Derenne JP, Milic-Emili J. Occlusion pressure as a measure of respiratory center output in conscious man. Respir Physiol. 1975 Mar;23(2):181-99. doi: 10.1016/0034-5687(75)90059-6. PMID 1144940
- [Result] Telias I, Damiani F, Brochard L. The airway occlusion pressure (P0.1) to monitor respiratory drive during mechanical ventilation: increasing awareness of a not-so-new problem. Intensive Care Med. 2018 Sep;44(9):1532-1535. doi: 10.1007/s00134-018-5045-8. Epub 2018 Jan 19. No abstract available. PMID 29350241
- [Result] Fossat G, Desmalles E, Courtes L, Fossat C, Boulain T. Cough Peak Flow Assessment Without Disconnection From the ICU Ventilator in Mechanically Ventilated Patients. Respir Care. 2023 Apr;68(4):470-477. doi: 10.4187/respcare.10412. Epub 2023 Mar 6. PMID 36878644
- [Result] Liang YR, Yang MC, Wu YK, Tzeng IS, Wu PY, Huang SY, Lan CC, Wu CP. Transitional Percentage of Minute Volume as a Novel Predictor of Weaning from Mechanical Ventilation in Patients with Chronic Respiratory Failure. Asian Nurs Res (Korean Soc Nurs Sci). 2020 Feb;14(1):30-35. doi: 10.1016/j.anr.2020.01.002. Epub 2020 Jan 22. PMID 31978600
- [Result] Souza LC, Lugon JR. The rapid shallow breathing index as a predictor of successful mechanical ventilation weaning: clinical utility when calculated from ventilator data. J Bras Pneumol. 2015 Nov-Dec;41(6):530-5. doi: 10.1590/S1806-37132015000000077. PMID 26785962
- [Result] Danaga AR, Gut AL, Antunes LC, Ferreira AL, Yamaguti FA, Christovan JC, Teixeira U, Guedes CA, Sasseron AB, Martin LC. Evaluation of the diagnostic performance and cut-off value for the rapid shallow breathing index in predicting extubation failure. J Bras Pneumol. 2009 Jun;35(6):541-7. doi: 10.1590/s1806-37132009000600007. English, Portuguese. PMID 19618034
- [Result] Camargo Barros Rocha DA, Marson FAL, Almeida CCB, Almeida Junior AA, Ribeiro JD. Association between oxygenation and ventilation indices with the time on invasive mechanical ventilation in infants. Pulmonology. 2018 Jul/Aug;24(4):241-249. doi: 10.1016/j.rppnen.2017.10.010. Epub 2018 Feb 2. PMID 29398628
- [Result] Paret G, Ziv T, Barzilai A, Ben-Abraham R, Vardi A, Manisterski Y, Barzilay Z. Ventilation index and outcome in children with acute respiratory distress syndrome. Pediatr Pulmonol. 1998 Aug;26(2):125-8. doi: 10.1002/(sici)1099-0496(199808)26:23.0.co;2-l. PMID 9727764
- [Result] Borman KR, Weigelt JA, Aurbakken CM. Guidelines for weaning from positive end-expiratory pressure in ventilated patients. Am J Surg. 1986 Dec;152(6):687-90. doi: 10.1016/0002-9610(86)90449-6. PMID 3538924
- [Result] Ramachandran V, Grap MJ, Sessler CN. Protocol-directed weaning: a process of continuous performance improvement. Crit Care. 2005 Apr;9(2):138-40. doi: 10.1186/cc3053. Epub 2005 Jan 28. PMID 15774063
- [Result] Walsh TS, Dodds S, McArdle F. Evaluation of simple criteria to predict successful weaning from mechanical ventilation in intensive care patients. Br J Anaesth. 2004 Jun;92(6):793-9. doi: 10.1093/bja/aeh139. Epub 2004 Apr 30. PMID 15121724
- [Result] Ely EW, Baker AM, Evans GW, Haponik EF. The prognostic significance of passing a daily screen of weaning parameters. Intensive Care Med. 1999 Jun;25(6):581-7. doi: 10.1007/s001340050906. PMID 10416909
- [Result] Shaw I, Gregory K. Acid-base balance: a review of normal physiology. BJA Educ. 2022 Oct;22(10):396-401. doi: 10.1016/j.bjae.2022.06.003. Epub 2022 Aug 18. No abstract available. PMID 36132879
- [Result] Hanley JA, McNeil BJ. The meaning and use of the area under a receiver operating characteristic (ROC) curve. Radiology. 1982 Apr;143(1):29-36. doi: 10.1148/radiology.143.1.7063747.
- [Result] Jiang JR, Yen SY, Chien JY, Liu HC, Wu YL, Chen CH. Predicting weaning and extubation outcomes in long-term mechanically ventilated patients using the modified Burns Wean Assessment Program scores. Respirology. 2014 May;19(4):576-82. doi: 10.1111/resp.12266. Epub 2014 Mar 24. PMID 24661343
- [Result] Nemer SN, Barbas CS, Caldeira JB, Carias TC, Santos RG, Almeida LC, Azeredo LM, Noe RA, Guimaraes BS, Souza PC. A new integrative weaning index of discontinuation from mechanical ventilation. Crit Care. 2009;13(5):R152. doi: 10.1186/cc8051. Epub 2009 Sep 22. PMID 19772625
- [Result] Burns SM, Fisher C, Earven Tribble SS, Lewis R, Merrel P, Conaway MR, Bleck TP. Multifactor clinical score and outcome of mechanical ventilation weaning trials: Burns Wean Assessment Program. Am J Crit Care. 2010 Sep;19(5):431-9. doi: 10.4037/ajcc2010273. PMID 20810418
- [Result] Menguy J, De Longeaux K, Bodenes L, Hourmant B, L'Her E. Defining predictors for successful mechanical ventilation weaning, using a data-mining process and artificial intelligence. Sci Rep. 2023 Nov 22;13(1):20483. doi: 10.1038/s41598-023-47452-7. PMID 37993526
- [Result] Baptistella AR, Sarmento FJ, da Silva KR, Baptistella SF, Taglietti M, Zuquello RA, Nunes Filho JR. Predictive factors of weaning from mechanical ventilation and extubation outcome: A systematic review. J Crit Care. 2018 Dec;48:56-62. doi: 10.1016/j.jcrc.2018.08.023. Epub 2018 Aug 20. PMID 30172034
- [Result] Baptistella AR, Mantelli LM, Matte L, Carvalho MEDRU, Fortunatti JA, Costa IZ, Haro FG, Turkot VLO, Baptistella SF, de Carvalho D, Nunes Filho JR. Prediction of extubation outcome in mechanically ventilated patients: Development and validation of the Extubation Predictive Score (ExPreS). PLoS One. 2021 Mar 18;16(3):e0248868. doi: 10.1371/journal.pone.0248868. eCollection 2021. PMID 33735250
- [Result] Fernandez MM, Gonzalez-Castro A, Magret M, Bouza MT, Ibanez M, Garcia C, Balerdi B, Mas A, Arauzo V, Anon JM, Ruiz F, Ferreres J, Tomas R, Alabert M, Tizon AI, Altaba S, Llamas N, Fernandez R. Reconnection to mechanical ventilation for 1 h after a successful spontaneous breathing trial reduces reintubation in critically ill patients: a multicenter randomized controlled trial. Intensive Care Med. 2017 Nov;43(11):1660-1667. doi: 10.1007/s00134-017-4911-0. Epub 2017 Sep 22. PMID 28936675
- [Result] Pham T, Heunks L, Bellani G, Madotto F, Aragao I, Beduneau G, Goligher EC, Grasselli G, Laake JH, Mancebo J, Penuelas O, Piquilloud L, Pesenti A, Wunsch H, van Haren F, Brochard L, Laffey JG; WEAN SAFE Investigators. Weaning from mechanical ventilation in intensive care units across 50 countries (WEAN SAFE): a multicentre, prospective, observational cohort study. Lancet Respir Med. 2023 May;11(5):465-476. doi: 10.1016/S2213-2600(22)00449-0. Epub 2023 Jan 21. PMID 36693401
- [Result] McConville JF, Kress JP. Weaning patients from the ventilator. N Engl J Med. 2012 Dec 6;367(23):2233-9. doi: 10.1056/NEJMra1203367. No abstract available. PMID 23215559
- [Result] Mabrouk AA, Mansour OF, El-Aziz AAA, Elhabashy MM, Alasdoudy AA (2015) Evaluation of some predictors for successful weaning from mechanical ventilation. Egyptian Journal of Chest Diseases and Tuberculosis 64:703-707
- [Result] Ouellette DR, Patel S, Girard TD, Morris PE, Schmidt GA, Truwit JD, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Kress JP. Liberation From Mechanical Ventilation in Critically Ill Adults: An Official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline: Inspiratory Pressure Augmentation During Spontaneous Breathing Trials, Protocols Minimizing Sedation, and Noninvasive Ventilation Immediately After Extubation. Chest. 2017 Jan;151(1):166-180. doi: 10.1016/j.chest.2016.10.036. Epub 2016 Nov 3. PMID 27818331
- [Result] Roberts KJ, Goodfellow LT, Battey-Muse CM, Hoerr CA, Carreon ML, Sorg ME, Glogowski J, Girard TD, MacIntyre NR, Hess DR. AARC Clinical Practice Guideline: Spontaneous Breathing Trials for Liberation From Adult Mechanical Ventilation. Respir Care. 2024 Jun 28;69(7):891-901. doi: 10.4187/respcare.11735. PMID 38443142
- [Result] Epstein SK. Weaning from ventilatory support. Curr Opin Crit Care. 2009 Feb;15(1):36-43. doi: 10.1097/MCC.0b013e3283220e07. PMID 19179869